CLINICAL TRIAL: NCT02260817
Title: Expanded Access to 11C Choline PET/CT and 11C Choline PET/MR for Staging of Recurrent Prostate Cancer With Comparison Study of CT and MR Modalities
Brief Title: Expanded Access to Diagnostic Imaging for Staging of Recurrent Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Isotopes, LLC d/b/a Zevacor Molecular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZM-CCH-40-PTL0114
Record Dates: First submitted 2014-08-04; First posted 2014-10-09 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate Cancer; 11C Choline; PET Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Expanded Access for 11C-Choline (Experimental): The key objective of this study is to provide expanded access to this drug product as currently defined under the reference listed drug as an investigational drug in geographical service areas where 11C-choline injection is not available.
  Patients entered into the study will undergo a 11C-choline PET CT scan and MRI scan. The 11C-choline PET CT and MRI images will be evaluated for evidence of metastatic prostate cancer. Patient data obtained in this arm of the study will not be further analyzed beyond that need for clinical diagnosis.
  Interventions: Drug: 11C-choline Injection
- 11C-Choline Comparison of Modalities (Experimental): 11C-choline injection is approved for use in conjunction with both CT and MR imaging modalities. This arm will attempt to determine which modality is most efficacious and under which conditions.
  Patients entered into the study will undergo imaging using GE's Trimodality Imaging System that combines PET, CT, and MR techniques to provide PET/CT and PET/MR fused images
  Interventions: Drug: 11C-choline Injection

INTERVENTIONS:
Drug: 11C-choline Injection — 1. Choline C11 Injection for PET/CT Imaging Protocol:
     * 15 - millicuries (mCi) 11C-choline IV Injection
     * PET images skull base to mid thigh with 3 min per bed position
     * Use of IV contrast based on American College of Radiology (ACR) IV contrast guidelines for a renal function screening protocol
     * Fusion of PET and CT images
  2. Choline C11 Injection for PET/MRI Whole Body Imaging Protocol:
     * No IV contrast
     * High resolution axial T2 prostate bed, axial Diffusion Weighted Image (DWI) pelvis, coronal T2 skull base to mid thighs
     * Fusion of coronal and PET images
  Other Names: CCH Injection, C11 Choline Injection

SUMMARY:
This Phase 3 study will target approximately 100 men over age 18 who have a biochemical relapse or other evidence of relapse of prostate cancer after primary treatment.

The purpose of this study is to:

A. Provide expanded access the drug 11C-choline.

B. Determine the performance characteristics (sensitivity, specificity, positive predictive value, negative predictive value) of 11C-choline PET/Computed Tomography (CT) and PET/Magnetic Resonance Imaging (MRI) in the detection of metastatic prostate cancer in patients with biochemical relapse of prostate cancer after primary treatment in a prospective manner.

C. Determine the optimal Prostate-Specific Antigen (PSA) trigger value in 11C-choline PET/CT and PET/MRI positive patients through a prospective study.

D. Determine factors that predict a confirmed positive 11C-choline PET/CT and PET/MRI using a multivariable analysis of clinical and pathologic data collected prospectively.

E. Compare the individual performance characteristics of 11C-choline PET/CT and 11C-choline PET/MRI and the combination of 11C-choline PET/CT and PET/MRI

Study Protocol:

1. Patients entered into the study will undergo a 11C-choline PET CT scan and MRI scan.
2. The CT and MRI images will be evaluated for evidence of metastatic prostate cancer.
3. The 11C-choline PET CT and MRI images will be evaluated for evidence of metastatic prostate cancer.
4. Evidence of metastasis on conventional imaging or 11C-choline PET will be confirmed with biopsy or surgical pathology when possible, or by response to treatment on subsequent imaging.
5. Rates of confirmed metastasis between conventional CT and MRI images will be compared with the 11C-choline PET CT and MRI images.
6. Upon conclusion of each imaging protocol, the referring physician will receive written documentation of the results. At this time, the patient will be considered off study and no further follow up is required.

DETAILED DESCRIPTION:
1. The first arm of this study serves to provide expanded access to 11C-choline injection as currently defined under the reference listed drug label as an investigational drug in geographical service areas where 11C-choline is not available. The second arm expands access as well but also attempts to determine the more effective imaging modality and conditions between PET/CT and PET/MR.
2. The study will consist of patients who have a biochemical relapse or other evidence of relapse after primary treatment. The first arm of the study is open to as many patients who elect to participate in the study that are over the age of 18 and have experienced a biochemical relapse of prostate cancer after primary treatment. The second arm will consist of patients who have been treated with radiation therapy, or androgen suppression and radiation therapy who have a PSA > 2 ng/mL higher than the nadir level. The nadir level in patients who have been treated with androgen suppression and radiation therapy is determined after the serum testosterone level has normalized. This study group will also consist of patients who have been treated with radical prostatectomy and who have a biochemical relapse defined as a PSA of 0.2 ng/mL confirmed at that level or higher on a subsequent PSA test 3 months later. This group may consist of men who have other clinical evidence of relapse such as a suspicious bone scan or CT scan regardless of PSA kinetics. Patients identified as potential subjects will be screened against the eligibility criteria as defined above in Section 5.1.
3. Informed consent will be obtained from all participants before any study related procedures are conducted. Each participant will be informed about the nature of the study, its purpose, and possible risks. Informed consent will be documented by using the written informed consent document approved by the local IRB at the Decatur Memorial Hospital.
4. At the time of referral, patients will be asked to bring their prior records as it pertains to their prostate cancer history. Data collected from outside records, such as radiographic studies, previous imaging studies and biopsies will be incorporated into the study record.
5. Abstracted data for the study record will include:

   1. Patient demographics such as age, race, and family history of prostate cancer
   2. Risk factors such as finasteride or dutasteride use, and environmental exposure (eg. Agent orange)
   3. Prostate exam results, most recent within last 90 days
   4. PSA test results, most current and past
   5. Past medical and surgical history
   6. Current medications
   7. Allergies
   8. Pathology reports
   9. Imaging reports
   10. Date of diagnosis
   11. Date(s) of biochemical relapse and coordinating PSA results. Once all records have been assessed for eligibility, an order for the 11C-choline PET CT scan and MRI scan will be requested from the referring physician and patient will be scheduled and given the appropriate prep instructions.
6. Both arms of the study will undergo a 11C-choline PET CT scan and MRI scan. The CT scan will be performed with intravenous contrast unless deemed unsafe by lab values. The CT and MRI images will be evaluated for evidence of metastatic prostate cancer. The 11C-choline PET CT and MRI images will be evaluated for evidence of metastatic prostate cancer. Unequivocal evidence of metastasis on both conventional imaging and 11C-choline PET will be considered a true positive. Evidence of metastasis on conventional imaging or 11C-choline PET will be confirmed with biopsy or surgical pathology when possible, or by response to treatment on subsequent imaging. If confirmation of metastasis is not achievable by biopsy or surgical pathology, then confirmation will be achieved with 11C-choline PET CT and MRI images obtained 3 months after treatment conclusion. Rates of confirmed metastasis between conventional CT and MRI images will be compared with the 11C-choline PET CT and MRI images.
7. Upon conclusion of each imaging protocol, the referring physician will receive written documentation of the results. At this time, the patient will be considered off study and no further follow up is required.

ELIGIBILITY:
Inclusion Criteria:

1. For biochemical relapse after primary treatment

   1. PSA > 0.2 ng/ml after radical prostatectomy confirmed at that level or higher on a subsequent test 3 months later
   2. PSA increase >2 ng/ml from nadir following radiation therapy
   3. PSA increase >2 ng/ml from nadir following radiation therapy plus androgen deprivation therapy with nadir defined with normalized testosterone level
   4. Two consecutive PSA increases from nadir level after androgen blockade or androgen suppression therapy
2. Kidney function with GFR > 60 mL/sec/1.73m2 and Creatinine < 1.7mg, collected within 90 days of planned scan

   1. if GFR is > or equal to 60 mL/sec/1.73m2, PET/CT will be completed with contrast
   2. if GFR is < 60 mL/sec/1.73m2, PET/CT will be completed without contrast
   3. if Creatinine is > than 1.7 mg, Radiology will follow ACR recommendations as outlined in department policy.
3. No known allergy to iodinated radiologic contrast media
4. Able to have MRI based on screening evaluation. If patient is found to be MRI incompatible, the 11C-choline PET/MRI portion of the study will not be completed. Please see the provided contact numbers for further options.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2

Exclusion Criteria:

1. ECOG Performance Status > 2.
2. Concurrent malignancy, i.e. colon cancer.
3. Treatment for another malignancy except superficial skin cancer within 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Tarter, M.D, Ph.D, Principal Investigator — Decatur Memorial Hospital
Locations (1):
- Decatur Memorial Hospital, Decatur, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 10/14 - 6/16, dosage and imaging only at Decatur Memorial Hospital in Decatur, IL.
Pre-assignment Details: No enrolled participants were excluded from either arm of the study prior to assignment.
Groups:
- 11C-choline for Staging of Recurrent Prostate Cancer: The key objective of this study is to provide expanded access to C11 Choline as an investigational drug in geographical service areas where it is not available.
  Patients entered into this arm of the study will undergo a 11C-choline PET CT scan and MRI scan. The 11C-choline PET CT and MRI images will be evaluated for evidence of metastatic prostate cancer. Patient data obtained in this arm will not be further analyzed beyond that need for clinical diagnosis.
- 11C-choline Comparison Study of CT and MR Modalities: 11C-choline injection is approved for use in conjunction with both CT and MR imaging modalities. This arm will attempt to determine which modality is most efficacious and under which conditions.
  Patients entered into the study will undergo imaging using GE's Trimodality Imaging System that combines PET, CT, and MR techniques to provide PET/CT and PET/MR fused images
  11C-choline Injection: 1. Choline C11 Injection for PET/CT Imaging Protocol:
  * 15 - millicuries (mCi) 11C-choline IV Injection
  * PET images skull base to mid thigh with 3 min per bed position
  * Use of IV contrast based on American College of Radiology (ACR) IV contrast guidelines for a renal function screening protocol
  * Fusion of PET and CT images
    2. Choline C11 Injection for PET/MRI Whole Body Imaging Protocol:
  * No IV contrast
  * High resolution axial T2 prostate bed, axial Diffusion Weighted Image (DWI) pelvis, coronal T2 skull base to mid thighs
  * Fusion of coronal and PET images
Period: Overall Study
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Started | 14 | 95
Completed | 14 | 58
Not Completed | 0 | 37
Not completed — Lost to Follow-up | 0 | 14
Not completed — Androgen deprivation therapy, no biopsy | 0 | 7
Not completed — Observation, no biopsy | 0 | 1
Not completed — Biopsy infeasible, ADT & rad. therapy | 0 | 1
Not completed — Protocol Violation | 0 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities | Total
Number analyzed (Participants) | 14 | 95 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 59 | 63
  >=65 years | 10 | 36 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 95 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 95 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 13 | 86 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 95 | 109

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Metastatic Prostate Cancer
Description: The CT and MRI images will be evaluated for evidence of metastatic prostate cancer. This Outcome is only measured for Arm 2 of this study.
  True Positive: True positives will consist of evidence of metastatic prostate cancer on conventional CT or MRI images or on 11C-choline PET/CT or MRI images confirmed with biopsy, surgical pathology, or by response to treatment with androgen suppression or other medical or radiation therapy.
  True Negative: True negatives will consist of negative images.
  False Positive: False positive will consist of evidence of metastatic prostate cancer on conventional CT or MRI images or on 11C-choline PET/CT or MRI images, but without corresponding confirmation from biopsy, surgical pathology or response to treatment.
  False Negative: False negative will consist of negative images, but with positive biopsy, surgical pathology or a response to treatment.
Time Frame: After 11C-choline PET CT scan and MRI scans, approximately 1 day. If surgery or response to treatment required to evaluate, approximately 1 to 3 months.
Population: Only those participants of Arm 2 not excluded due to reasons listed in Population Flow were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
Participants
  True Positive | 0 | 36
  True Negative | 0 | 10
  False Positive | 0 | 11
  False Negative | 0 | 1

2. Primary Outcome: Sensitivity of 11C Choline PET Imaging Scans
Description: The results of the population's 11C-choline PET CT scans and MRI scans will be evaluated for imaging sensitivity.
  Sensitivity of 11C-choline PET/CT and MRI will be calculated as True Positive / (True Positive + False Negative).
  This Outcome is only measured for Arm 2 of this study.
Time Frame: Approximately 1 day post-scan for patient results
Population: Only those participants of Arm 2 not excluded due to reasons listed in Population Flow were analyzed for this outcome.
Measure: Number; unit: % of correctly identified positives
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
% of correctly identified positives |  | 97.29

3. Primary Outcome: Specificity of 11C Choline PET Imaging Scans
Description: The results of the population's 11C-choline PET CT scans and MRI scans will be evaluated for imaging specificity.
  Specificity of 11C-choline PET/CT and MRI will be calculated as True Negative / (True Negative + False Positive).
  This Outcome is only measured and reported for Arm 2.
Time Frame: Approximately 1 day post-scan for patient results
Population: Only those participants of Arm 2 not excluded due to reasons listed in Population Flow were analyzed for this outcome.
Measure: Number; unit: % correctly identified negatives
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
% correctly identified negatives |  | 47.61

4. Primary Outcome: Positive Predictive Value (PPV) of 11C Choline PET Imaging Scans
Description: The results of the population's 11C-choline PET CT scans and MRI scans will be evaluated for the images' positive predictive value.
  Positive Predictive Value of 11C-choline PET/CT and MRI will be calculated as True Positive / (True Positive + False Positive).
  This Outcome is only measured for Arm 2.
Time Frame: Approximately 1 day post-scan for patient results
Population: Only those participants of Arm 2 not excluded due to reasons listed in Population Flow were analyzed for this outcome.
Measure: Number; unit: Probability of disease (%)
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
Probability of disease (%) |  | 76.59

5. Primary Outcome: Negative Predictive Value (NPV) of 11C Choline PET Imaging Scans
Description: The results of the population's 11C-choline PET CT scans and MRI scans will be evaluated for the images' negative predictive value.
  Negative Predictive Value of 11C-choline PET/CT and MRI will be calculated as True Negative / (True Negative + False Negative).
  This Outcome is only measured for Arm 2.
Time Frame: Approximately 1 day post-scan for patient results
Population: Only those participants of Arm 2 not excluded due to reasons listed in Population Flow were analyzed for this outcome.
Measure: Number; unit: Probability of being disease-free (%)
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
Probability of being disease-free (%) |  | 90.90

6. Primary Outcome: Count of Participants With Positive or Negative PET, CT, or MRI Modalities Resulting in Prostate Cancer (PCa) Confirmation
Description: Comparison of the results of participants' imaging modalities and whether those imaging modalities resulted in confirmation of Prostate Cancer (PCa). This Outcome is only measured for Arm 2.
Time Frame: Approximately 1 day post-scan for patient results
Population: This population only includes those Arm 2 participants with positive PET imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 36
Participants
  Positive PET, Negative CT, Negative MRI |  | 11
  Positive PET, Positive CT, Negative MRI |  | 6
  Positive PET, Negative CT, Positive MRI |  | 11
  Positive PET, Positive CT, Positive MRI |  | 8

7. Secondary Outcome: Median Age at Primary Treatment
Description: The median age at primary treatment for Arm 2 participants.
Time Frame: The participants' age at primary treatment was collected upon study enrollment (approximately 1 week into study)
Population: Only Arm 2 participants' data was collected.
Measure: Median (Full Range); unit: years
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
years |  | 63 [48 to 82]

8. Secondary Outcome: Median PSA at Diagnosis of Arm 2 Participants
Description: The Prostate-Specific Antigen (PSA) measurement of participants at their original prostate cancer diagnosis was collected at entry to this trial. It is reported as nanograms of PSA per milliliter (ng/mL) of blood. The Median of all reported PSAs is reported here.
Time Frame: The participants' primary PSA at diagnosis was collected upon study enrollment (approximately 1 week into study)
Population: Only Arm 2 participants' data was collected. *Note: 4 participants' PSA was not reported.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 54
ng/ml |  | 13.07 [1.29 to 105]

9. Secondary Outcome: Clinical T (cT) Stage of Arm 2 Participants
Description: An accounting of the approximate clinical (pre-treatment) stage for the Arm 2 participants. Clinical staging is based on the results of tests done before surgery.
  T1: PC is too small to be seen on a scan or felt during prostate examination
  T1a: PC is in < 5% of removed tissue
  T1b: PC is in > 5% or more of removed tissue
  T1c: PC is found by biopsy
  T2: PC is completely inside prostate
  T2a: PC is in only half of one side of prostate
  T2b: PC is in more than half of one side of prostate, but not both sides
  T2c: PC is in both sides but is still inside prostate
  T3: PC has broken through the capsule of prostate
  T3a: PC has broken through the capsule of prostate
  T3b: PC has spread into seminal vesicles
  T4: PC has spread into other nearby body organs
Time Frame: The participants' clinical stage data was collected upon study enrollment (approximately 1 week into study)
Population: Only data from Arm 2 participants' was collected. Note: Clinical Staging for 4 participants was not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 54
Participants
  cT Stage: T1c | 0 | 34
  cT Stage: T2 | 0 | 20

10. Secondary Outcome: Median Primary Biopsy Gleason Score of Arm 2 Participants
Description: The median primary Biopsy Gleason Score for the Arm 2 participants' will be reported.
  The Gleason Score is the grading system used to determine the aggressiveness of prostate cancer. Typical Gleason Scores range from 6-10. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly.
  Gleason scores 2-4 are typically found in smaller tumors located in the transitional zone (around the urethra).
  The majority of treatable/treated cancers are of Gleason scores 5 - 7 and are detected due to biopsy after abnormal digital rectal exam or prostate specific antigen evaluation. The cancer is typically located in the peripheral zone usually the posterior portion.
  Tumors with Gleason scores 8-10 tend to be advanced neoplasms that are unlikely to be cured.
Time Frame: The participants' primary Biopsy Gleason Score data was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 Participants. Note: Biopsy Gleason Grade was not reported for 1 participant.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 57
units on a scale |  | 7 [5 to 9]

11. Secondary Outcome: Primary Treatment Modality of Arm 2 Participants
Description: An accounting of the primary treatment modalities undergone by the participants in Arm 2 prior to their involvement in the trial will be reported.
  Modalities reported below are:
  Androgen Deprivation Therapy (ADT) External Beam Radiation Therapy (EBRT) Brachytherapy Cryoablation Cystoprostatectomy Intensity-Modulated Radiation Therapy (IMRT) Radical Prostatectomy (RP)
Time Frame: The participants' primary treatment data was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
Participants
  ADT |  | 1
  ADT + Brachytherapy |  | 1
  ADT + EBRT + Brachytherapy |  | 2
  Brachytherapy |  | 4
  Brachytherapy + EBRT |  | 1
  Cystoprostratectomy |  | 1
  EBRT |  | 10
  EBRT + ADT |  | 3
  IMRT |  | 1
  RP |  | 34

12. Secondary Outcome: Pathological Stage (pT) of Prostate Cancer (PC) of Arm 2 Participants
Description: The pathological stage of PC at primary diagnosis for Arm 2 participants was collected. pT is based on how different from normal the cells in samples of tissue recovered from surgery look under a microscope.
  T1: PC is too small to be seen on a scan or felt during prostate examination
  T1a: PC is in < 5% of removed tissue
  T1b: PC is in > 5% or more of removed tissue
  T1c: PC is found by biopsy
  T2: PC is completely inside prostate
  T2a: PC is in only half of one side of prostate
  T2b: PC is in more than half of one side of prostate, but not both sides
  T2c: PC is in both sides but is still inside prostate
  T3: PC has broken through the capsule of prostate
  T3a: PC has broken through the capsule of prostate
  T3b: PC has spread into seminal vesicles
  T4: PC has spread into other nearby body organs
Time Frame: The participants' primary pathological staging data was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 participants. Note: Pathological Stage data not collected for 26 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 32
Participants
  pT2a |  | 1
  pT2c |  | 14
  pT3a |  | 9
  pT3b |  | 8

13. Secondary Outcome: Primary Surgical Margins of Arm 2 Participants
Description: A census of the primary surgical margins of participants in Arm 2 will reported.
  The surgical margins are the set of surfaces that were cut by the surgeon in order to remove the specimen from the body.
  Positive Margin: surgical margins with disease present. Negative Margin: surgical margins with no disease present.
Time Frame: The participants' primary surgical margins data was collected upon study enrollment (approximately 1 week into study)
Population: Only data for Arm 2 participants was collected. Note: Primary Surgical Margins were not collected for 26 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 32
Participants
  Negative Surgical Margins |  | 13
  Positive Surgical Margins |  | 19

14. Secondary Outcome: Primary Positive Lymph Node Ratio of Arm 2 Participants
Description: A census of the positive lymph node ratio, defined as ratio of positive lymph nodes to all lymph nodes removed, for the participants of Arm 2 will be reported.
  The N refers to the the number of nearby lymph nodes that have cancer. NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
Time Frame: The participants' primary positive lymph note ratio was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 participants. Note: Primary Positive Lymph Node Ratio was not collected for 26 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 32
Participants
  NX |  | 3
  N0 |  | 25
  N1 |  | 4

15. Secondary Outcome: Additional Treatment and Type for Arm 2 Participants
Description: A census of the additional treatments undergone by participants prior to enrollment in the study, if undergone, for the participants of Arm 2 will be reported.
  None Androgen Deprivation Therapy (ADT) Radiation Therapy (RT) Electron Beam Radiation Therapy (EBRT) Lycopene (herbal treatment) Salvage Radiation Therapy (RT) Salvage Radical Prostatectomy (RP) Adjuvant Radiation Therapy (RT) Bilateral Pelvis Lymph Node Dissection
Time Frame: The participants' additional primary treatment data was collected upon study enrollment (approximately 1 week into study)
Population: only data from Arm 2 Participants is collected. Note: Additional Treatment was not reported for 1 participant.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 57
Participants
  Adjuvant RT |  | 3
  ADT |  | 11
  Bilateral Pelvis Lymph Node Dissection |  | 1
  EBRT |  | 1
  Lycopene |  | 1
  None |  | 31
  Salvage RP |  | 1
  Salvage RT |  | 5
  Salvage RT + ADT |  | 3

16. Secondary Outcome: Median Months to Biochemical Relapse of Arm 2 Participants
Description: The median of the Arm 2 participants' data between initial treatment and biochemical relapse, occurring prior to study enrollment, measured in months, will be reported.
Time Frame: The participants' biochemical relapse data was collected upon study enrollment (approximately 1 week into study)
Population: only data from Arm 2 participants is collected. Note: Biochemical Relapse Data was not collected for 2 participants.
Measure: Median (Full Range); unit: months
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 56
months |  | 40 [2 to 197]

17. Secondary Outcome: Median Age of Arm 2 Participant at PET Imaging
Description: The median age (at time of study) of participants of Arm 2 will be reported in years.
Time Frame: The participants' age at study entry was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 participants is reported.
Measure: Median (Full Range); unit: years
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
years |  | 69 [50 to 86]

18. Secondary Outcome: Median PSA of Arm 2 Participant at PET Imaging
Description: The median of the PSA of Arm 2 participants at study entry will be reported as nanograms of PSA per milliliter (ng/mL) of blood
Time Frame: The participants' PSA was collected upon study enrollment (approximately 1 week into study)
Population: only data collected for Arm 2 participants.
Measure: Median (Full Range); unit: ng/ml of blood
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 58
ng/ml of blood |  | 3.58 [0.24 to 107.9]

19. Secondary Outcome: Median PSA Doubling Time of Arm 2 Participants at PET Imaging
Description: The median of the time, measured in months that an Arm 2 participant's PSA has doubled from initial diagnosis to PSA measured at study enrollment.
Time Frame: The participants' PSA doubling time was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 participants is reported. Note: PSA doubling time (in months) was not collected for 3 participants.
Measure: Median (Full Range); unit: months
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 55
months |  | 4.91 [0 to 35.3]

20. Secondary Outcome: Median PSA Velocity of Arm 2 Participants at PET Imaging
Description: The median PSA velocity (measured in ng/mL/month) of the Arm 2 participants will be reported.
Time Frame: The participants' PSA velocity was collected upon study enrollment (approximately 1 week into study)
Population: Only data collected from Arm 2 participants is reported. Note: PSA velocity was not collected for 3 participants.
Measure: Median (Full Range); unit: ng/mL/month
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 55
ng/mL/month |  | 0.09 [0 to 2.42]

21. Secondary Outcome: ADT (Androgen Deprivation Therapy) in Participant at PET Imaging
Description: An accounting of whether the participants of Arm 2 have undergone androgen deprivation therapy (ADT).
Time Frame: The participants' participation in ADT was collected upon study enrollment (approximately 1 week into study)
Population: Only the Arm 2 participants data is reported. Note: ADT information was not collected for 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
Number analyzed (Participants) | 0 | 56
Participants
  No ADT received |  | 48
  ADT received |  | 8

ADVERSE EVENTS:
Time Frame: Participants were monitored throughout the imaging process during the administration of the imaging agents and immediately thereafter. They were contacted within 1 day after the scan for assessment.
Description: Adverse Events were assessed per the standard Adverse Events definition. Patients were contacted by telephone 24 hours post-C11 Choline PET scan for any follow-up concerns and were also told to report any immediate or additional concerns.
Arm/Group | 11C-choline for Staging of Recurrent Prostate Cancer | 11C-choline Comparison Study of CT and MR Modalities
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/95
Other Adverse Events (participants affected / at risk) | 0/14 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02260817/Prot_SAP_000.pdf